CLINICAL TRIAL: NCT05069922
Title: Randomized Trial of Fresh Frozen Plasma Versus Albumin in Acute Burn Resuscitation
Acronym: FFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-3710; CDMRP-MB200032 (Other: USAMRAA)
Record Dates: First submitted 2021-09-27; First posted 2021-10-06 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Burns
Keywords: Burn resuscitation
MeSH Terms: conditions — Burns | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh Frozen Plasma (Active Comparator): At 6-8 hours, Initiate FFP infusion
  Interventions: Other: Fresh Frozen Plasma
- Albumin (Active Comparator): At 7 hours, Initiate 5% Albumin infusion
  Interventions: Other: Fresh Frozen Plasma

INTERVENTIONS:
Other: Fresh Frozen Plasma — Fresh Frozen Plasma
  Other Names: Albumin

SUMMARY:
The investigators propose a prospective randomized trial to study fresh frozen plasma (FFP) versus albumin to determine the optimal colloid in burn resuscitations. This work addresses both FY20 focus areas, prolonged field care (PFC) and en route care, along with mitigating secondary effects of acute intervention, such as prevention of over resuscitation. Future military conflicts anticipate more extensive burn and blast injuries, and delayed evacuation. Therefore, the direct comparison of colloids used in burn resuscitation is critical to advancing battlefield medicine. Specifically, this work will provide the foundation for the use of freeze-dried plasma (FDP) in burn care by medical responders in PFC and en route care scenarios. The investigators hypothesize that FFP administration, and later FDP, in burn resuscitation is as safe as albumin, and more efficacious, in both reducing the total volume of fluid required in acute burn resuscitation and correcting burn endotheliopathy.

DETAILED DESCRIPTION:
Specific Aim 1: The investigators will evaluate the total fluids administered in FFP (intervention) and albumin (control) groups. The investigators propose that the FFP group will require less total fluids administered.

Specific Aim 2:The investigators will determine overall complication rates (pulmonary complications, ARDS, ACS, over-resuscitation) in the FFP (intervention) and albumin (control) administration groups. The investigators propose FFP administration will reduce the frequency of these complications.

Specific Aim 3: The investigators will characterize the effects of FFP and albumin administration on endothelial dysfunction in major burns. We will measure glycocalyx degradation products (e.g. syndecan-1, glycosaminoglycans) in the serum. The investigators project FFP will mitigate GDP better than albumin.

ELIGIBILITY:
Inclusion Criteria:

* adult thermal injury patients aged 2:18 years old with burns ->20% TBSA seen at UCH Burn Center within 8 hours of burn injury

Exclusion Criteria:

* Pregnant patients, prisoners, Jehovah's Witness/inability to receive human blood product/component therapy, electrical injury, chemical injury, friction/shear injury, anticipated death within 48 hours of admission, delayed intervention (>8 hours post burn), history of renal failure requiring dialysis, Stage IV or V chronic kidney disease, coagulopathy (admission INR >2.5), cirrhosis (Childs B,C), concomitant life threatening traumatic injuries, receiving blood product transfusion for another reason, inability to obtain consent from patient or legally authorized representative.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Total volume of fluid administered in 24 hours in each group (FFP or albumin), measured as mL/kg/%TBSA burned. | 3 years
  Total volume

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Data will be compiled and shared with Department of Defense